CLINICAL TRIAL: NCT07245186
Title: Exploring Approaches for Proactive Health in People With Kidney Function Decline: Insights From a Prospective Cohort Study
Brief Title: Strategies for Proactive Health in People With Kidney Function Decline
Status: Enrolling by invitation | Type: Observational
Sponsor: Huashan Hospital (Other)
Collaborators: Jingan District Central Hospital of Shanghai (Jingan Branch of Huashan Hospital Affiliated to Fudan University) (Unknown); Shanghai Changfeng community Healthcare center, Putuo, Shanghai, China (Unknown)
Responsible Party: Principal Investigator, Chen Jing, Professor, Huashan Hospital
Other Study IDs: KY2023-973
Record Dates: First submitted 2025-11-16; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Renal Insufficiency,Chronic; Dietary Intake Patterns; Malnutrition; Frailty; Cognitive Dysfunction; CKD-MBD - Chronic Kidney Disease Mineral and Bone Disorder
Keywords: Kidney Function Decline; Nutritional Intake; Dietary Assessment; Health Outcomes; Cohort Study
MeSH Terms: conditions — Renal Insufficiency, Chronic; Malnutrition; Frailty; Cognitive Dysfunction; Chronic Kidney Disease-Mineral and Bone Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with renal function decline (non-dialysis cohort): This is a multi-center prospective cohort study led by Huashan Hospital, Fudan University, with collaboration from several other hospitals. The study aims to recruit at least1800 participants, primarily older adults, with varying degrees of kidney function decline, with enrollment ongoing from January 2021 to December 2029.
  Participants undergo baseline assessments, including dietary intake surveys, biochemical and metabolic testing, body composition analysis, and clinical evaluations. Follow-up assessments are conducted at predetermined intervals to monitor kidney function, cardiovascular health, metabolic status, and overall well-being.
  This cohort provides a structured platform for long-term observational research on the relationship between nutrition, metabolism, and health outcomes in aging populations. The findings will support the development of precision nutrition strategies and proactive aging health management.

SUMMARY:
This prospective cohort study aims to investigate how kidney function decline affects multiple body systems and how personalized nutrition can help maintain health and slow disease progression. About 1,800 adults with reduced kidney function but not on dialysis will be followed over time at Huashan Hospital, Fudan University. The study will collect information on nutrition, heart and bone health, cognition, and daily functioning through hospital records and a patient mobile app. The goal is to understand the links between nutrition, metabolism, and organ function, and to develop integrated strategies for early prevention and management of chronic kidney disease.

DETAILED DESCRIPTION:
Kidney function often declines gradually with age or chronic conditions, even before chronic kidney disease is formally diagnosed. This decline can disturb the body's overall balance, leading to changes in heart and blood vessel health, bone metabolism, muscle strength, and cognitive performance. Nutrition and metabolism play central roles in these processes, but how they interact during kidney function decline remains unclear.

This prospective cohort study, conducted at Huashan Hospital, Fudan University, aims to understand the multisystem changes that occur during kidney function decline and to explore how individualized, nutrition-integrated management can help maintain health and slow disease progression. Approximately 1,800 adults with an estimated glomerular filtration rate (eGFR) below 90 mL/min/1.73 m² and not receiving dialysis will be enrolled and followed for up to ten years.

Comprehensive information on participants' diet, biochemical markers, heart and bone health, cognition, and physical function will be collected through hospital systems and a mobile nutrition management app. The study seeks to identify how nutritional status and metabolic adaptation relate to outcomes such as kidney function decline, cardiovascular disease, frailty, and cognitive impairment. Findings from this research will help develop an integrated, multidisciplinary approach to prevent complications and improve the overall health and quality of life of people with reduced kidney function.

ELIGIBILITY:
Inclusion Criteria:

1. Non-dialysis patients with chronic kidney disease (CKD) stages 1-5.
2. Aged 18 to 90 years, no restriction on gender.
3. Sufficient health literacy or a family member with adequate literacy to comply with dietary diary recording and other study procedures.
4. Stable primary disease of CKD at the time of enrollment.

Exclusion Criteria:

1. Patients with malignancies, severe cardiovascular diseases, osteoporosis, or severe hematological disorders.
2. Active infections (CRP >10 mg/L) or current use of nephrotoxic drugs.
3. Limb paralysis or amputation.
4. Use of immunosuppressants (cyclosporine, tacrolimus) within the past 3 months or steroid therapy equivalent to prednisone >10 mg/day.
5. Severe gastrointestinal diseases affecting nutrient absorption.
6. Participation in other diet- or drug-related clinical studies within the past month or ongoing.
7. Any other condition deemed inappropriate for participation by the investigators.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 years or older with reduced kidney function (eGFR < 90 mL/min/1.73 m²) who are not receiving dialysis. Participants are recruited from outpatient clinics at Huashan Hospital, Fudan University.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2029-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Rapid decline in renal function | eGFR will be measured at baseline and at 1 month, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 30 months, and 36 months after enrollment, and subsequently every 6 months thereafter up to 10 years of follow-up.
  The primary outcome is the occurrence of a rapid decline in kidney function, defined as a ≥40% decrease in estimated glomerular filtration rate (eGFR) from baseline during the follow-up period. eGFR will be calculated using the CKD-EPI formula based on serum creatinine measurements obtained during scheduled clinical visits.

SECONDARY OUTCOMES:
End-Stage Renal Disease (ESRD) | Assessed at baseline and every follow-up visit (1 month, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 30 months, 36 months, and every 6 months thereafter up to 10 years).
  The occurrence of end-stage renal disease (ESRD), defined as initiation of renal replacement therapy, including maintenance dialysis (hemodialysis or peritoneal dialysis) or receipt of kidney transplantation. ESRD events will be confirmed through clinical records and verified by treating nephrologists.
Incidence of Cardiovascular Events | Evaluated at baseline, at 6 months, at 1 year, and annually thereafter up to 10 years.
  Composite incidence of cardiovascular and cerebrovascular events, including coronary artery disease, cardiac arrhythmia, stroke, heart failure, and sudden cardiac death. All events will be confirmed through medical records, imaging examinations, and classified according to international diagnostic standards.
All-Cause Mortality | Assessed at baseline and every follow-up visit (1 month, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 30 months, 36 months, and every 6 months thereafter up to 10 years).
  All-cause mortality includes death due to any cause, with a specific focus on deaths related to kidney disease progression and its complications, particularly cardiovascular disease, infections, and other related conditions. Deaths will be verified through medical records and official documentation.
Cognitive Impairment | Evaluated at baseline, 12 months, 24 months, 36 months, and every 2 years thereafter up to 10 years.
  Cognitive function will be assessed using the Mini-Mental State Examination (MMSE) and the Montreal Cognitive Assessment (MoCA). MMSE scores <27 and MoCA scores <26 indicate cognitive impairment. Severity will be classified as mild, moderate, or severe based on standardized score ranges and adjusted for education level.
Frailty | Measured at baseline, 12 months, 24 months, 36 months, and every 2 years thereafter up to 10 years.
  Frailty will be determined using the Fried frailty phenotype, defined by the presence of three or more of the following criteria: unintentional weight loss (≥4.5 kg or ≥5% within one year), self-reported exhaustion, weakness (grip strength adjusted for sex and BMI), slow walking speed (adjusted for sex and height), and low physical activity level assessed by the Minnesota Leisure Time Activity Questionnaire.
Malnutrition and Protein-Energy Wasting (PEW) | Assessed at baseline, 6 months, 12 months, 24 months, 36 months, and every 12 months thereafter up to 10 years.
  Nutritional status will be evaluated according to both the GLIM criteria and the ISRNM definition of protein-energy wasting (PEW). GLIM diagnosis requires at least one phenotypic criterion (unintentional weight loss, low BMI, or reduced muscle mass by BIA or ultrasound) and one etiologic criterion (reduced food intake/absorption or disease burden/inflammation). PEW is defined by abnormalities in at least three of four domains: biochemical markers, body composition, muscle mass, and dietary intake, according to ISRNM standards.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Chen, PhD, MD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan hospital, Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No